CLINICAL TRIAL: NCT03093389
Title: A Double-blind, Randomised, Placebo-controlled, Rising Multiple-dose Study to Investigate the Tolerability and Steady-state Pharmacokinetics of BIA 6-512 (Trans-resveratrol) in Healthy Volunteers
Brief Title: Tolerability and Steady-state Pharmacokinetics of BIA 6-512
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-6512-103
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BIA 6-512 25 mg or Placebo (Experimental): 1 capsule of BIA 6-512 25 mg or 1 capsule of placebo.
  Interventions: Drug: BIA 6-512; Drug: Placebo
- BIA 6-512 50 mg or Placebo (Experimental): 1 capsule of BIA 6-512 50 mg or 1 capsule of placebo.
  Interventions: Drug: BIA 6-512; Drug: Placebo
- BIA 6-512 100 mg or Placebo (Experimental): 1 capsule of BIA 6-512 100 mg or 1 capsule of placebo.
  Interventions: Drug: BIA 6-512; Drug: Placebo
- BIA 6-512 150 mg or Placebo (Experimental): 1 capsule of BIA 6-512 150 mg or 1 capsule of placebo.
  Interventions: Drug: BIA 6-512; Drug: Placebo

INTERVENTIONS:
Drug: BIA 6-512 — The investigational products consisted of capsules containing BIA 6-512 25 mg, 50 mg, 100 mg and 150 mg. Products were administered orally, with approximately 240 mL of water in case of Doses 1 and 13, and at least 150 mL of water in case of Doses 2 to 12. First dose (Dose 1) and last dose (Dose 13) were administered in fasting of at least 8 hours and subject remained fasted until to 2.5 h post-dose. Meals were not served within 1 hour prior and 1 hour after investigational product administration in Doses 2 to 12
  Other Names: Trans-resveratrol
Drug: Placebo — Matching placebo capsules

SUMMARY:
To investigate the tolerability and safety of four multiple-dose regimens of BIA 6-512 (25 mg, 50 mg, 100 mg, and 150 mg 6 times daily) in healthy volunteers and to characterise the steady-state pharmacokinetic profiles of BIA 6-512 (25 mg, 50 mg, 100 mg, and 150 mg 6 times daily) in healthy volunteers.

DETAILED DESCRIPTION:
Single-centre, double-blind, randomised, placebo-controlled study of four multiple-rising doses in four sequential groups of 10 healthy volunteers each. Eligible subjects were admitted to the UFH on the day (Day 0) prior to receiving the first dose of study medication. On the morning of the next day (Day 1), subjects started receiving BIA 6-512/Placebo at 4 h intervals (6 times/day) for 48 h (13 investigational product administrations, in total). Subjects remained confined in the UFH from admission (Day 0) until at least 24 h post last dose (Day 4); then, they were discharged and were requested to return for the follow-up visit. At given time-points, subjects were submitted to vital signs recording, brief neurological examination, and 12-lead ECG. Blood samples for plasma drug assays were taken at the following times: Dose 1: pre-dose and ¼, ½, ¾, 1, 1½, 2, and 3 hours post-dose; Doses 2, 3, 4, 5, 7, 8, 9, 10, 11: pre-dose; Dose 13: pre-dose and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Subjects who had clinical laboratory test results clinically acceptable at screening and admission.
* Subjects who had negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening.
* Subjects who had a negative screen for alcohol and drugs of abuse at screening and admission.
* Subjects who were non-smokers or who smoke ≤ 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.
* (If female) She had a negative urine pregnancy test at screening and admission.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria, or
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant drug or food hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 21 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening or admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used medicines within 2 weeks of first admission that, in the opinion of the investigator, may affect the safety or other study assessments.
* Subjects who had used any investigational drug or participated in any clinical trial within 2 months of their admission.
* Subjects who had donated or received any blood or blood products within the previous 2 months prior to screening.
* Subjects who were vegetarians, vegans or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an approved effective contraceptive method (double-barrier, intra-uterine device or abstinence) or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-05-11 (Actual); Primary Completion 2005-07-29 (Actual); Study Completion 2005-07-29 (Actual)

PRIMARY OUTCOMES:
Cmax - the maximum plasma concentration - first dose (dose 1) | Dose 1: pre-dose and ¼, ½, ¾, 1, 1½, 2, and 3 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the first dose (Dose 1)
tmax - the time of occurrence of Cmax - first dose (dose 1) | Dose 1: pre-dose and ¼, ½, ¾, 1, 1½, 2, and 3 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the first dose (Dose 1)
AUC0-t - the area under the plasma concentration-time curve from time zero to the last sampling time at which concentrations are at or above the limit of quantification, calculated by the linear trapezoidal rule - first dose (dose 1) | Dose 1: pre-dose and ¼, ½, ¾, 1, 1½, 2, and 3 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the first dose (Dose 1)
AUC0-τ - the area under the plasma concentration versus time curve over the dosing interval (4 h), calculated by the linear trapezoidal rule - first dose (dose 1) | Dose 1: pre-dose and ¼, ½, ¾, 1, 1½, 2, and 3 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the first dose (Dose 1)
AUC0-¥ - the area under the plasma concentration versus time curve from time zero to infinity, calculated from AUC0-t + (Clast/lz), where Clast is the last quantifiable concentration and lz the apparent terminal rate constant - first dose (dose 1) | Dose 1: pre-dose and ¼, ½, ¾, 1, 1½, 2, and 3 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the first dose (Dose 1)
t½ - the apparent elimination half-life, calculated from ln 2/lz - first dose (dose 1) | Dose 1: pre-dose and ¼, ½, ¾, 1, 1½, 2, and 3 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the first dose (Dose 1)
Cmax - the maximum plasma concentration - last dose (dose 13) | Dose 13: pre-dose and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the last dose (Dose 13)
tmax - the time of occurrence of Cmax - last dose (dose 13) | Dose 13: pre-dose and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the last dose (Dose 13)
AUC0-t - the area under the plasma concentration-time curve from time zero to the last sampling time at which concentrations are at or above the limit of quantification, calculated by the linear trapezoidal rule - last dose (dose 13) | Dose 13: pre-dose and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the last dose (Dose 13)
AUC0-τ - the area under the plasma concentration versus time curve over the dosing interval (4 h), calculated by the linear trapezoidal rule - last dose (dose 13) | Dose 13: pre-dose and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the last dose (Dose 13)
AUC0-¥ - the area under the plasma concentration versus time curve from time zero to infinity, calculated from AUC0-t + (Clast/lz), where Clast is the last quantifiable concentration and lz the apparent terminal rate constant - last dose (dose 13) | Dose 13: pre-dose and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the last dose (Dose 13)
t½ - the apparent elimination half-life, calculated from ln 2/lz - last dose (dose 13) | Dose 13: pre-dose and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  BIA 6-512 pharmacokinetic parameters following the last dose (Dose 13)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit (UFH) - BIAL - Portela & Cª, SA, S. Mamede Do Coronado, Portugal

IPD SHARING:
Plan to Share IPD: Undecided